CLINICAL TRIAL: NCT07271615
Title: Preoperative Stellate Ganglion Block Reduce the Incidence of Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting: A Prospective, Randomized Controlled Pilot Trial
Brief Title: Effect of Preoperative Stellate Ganglion Block on Postoperative Atrial Fibrillation After Coronary Artery Bypass Grafting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, MD，phD, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20250716
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Adult Patients Undergoing CABG

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group（C group） (No Intervention): the best available treatment without block (usual care)
- Stellate Ganglion Block（S group） (Other): Ultrasound-guided stellate ganglion block with ropivacaine
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Ultrasound-guided stellate ganglion block with ropivacaine
  Arms: Stellate Ganglion Block（S group）

SUMMARY:
The primary objective of this study is to determine the feasibility of preoperative stellate ganglion block in reducing the incidence of postoperative atrial fibrillation in patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* undergoing CABG
* Provide informed consent

Exclusion Criteria:

* History of prior cardiac surgery or atrial fibrillation ablation;
* Emergency coronary artery bypass grafting (CABG);
* Concomitant cardiac procedures (e.g., congenital heart disease repair, left ventricular reconstruction, valve surgery, or aortic surgery);
* Critical preoperative status requiring mechanical or pharmacological support before CABG;
* Left ventricular ejection fraction (LVEF) <35%;
* History of atrial fibrillation (defined as a supraventricular tachyarrhythmia characterized by rapid and irregular atrial electrical activity);
* Significant mitral valve disease (mitral valve area <1.5 cm² or regurgitant jet area <4 cm²), significant aortic valve disease (valve area <1.5 cm² or regurgitant jet-to-left ventricular outflow tract ratio >25%);
* Severe left atrial enlargement (left atrial anteroposterior diameter >55 mm);
* Poorly controlled hyperthyroidism;
* Conditions requiring radiotherapy, chemotherapy, or long-term hormonal therapy;
* Patients with known clinical contraindications to stellate ganglion block (SGB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative atrial fibrillation（POAF） | within 7 days postoperatively

SECONDARY OUTCOMES:
cumulative time spent in postoperative atrial fibrillation | within 7 days postoperatively
the need for antiarrhythmic medications to treat postoperative atrial fibrillation | within 7 days postoperatively
the need for systemic anticoagulation due to postoperative atrial fibrillation | within 7 days postoperatively
the need for postoperative electrical cardioversion | within 7 days postoperatively
the duration of postoperative in-hospital stay | duration of postoperative hospital stay
number of POAF | within 7 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China